CLINICAL TRIAL: NCT03094338
Title: A Stress Survey in Nurse Anesthetist Students
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Supaporn Laotaweesuk, Nurse anesthetist, Siriraj Hospital
Other Study IDs: Si 099/2017
Record Dates: First submitted 2017-03-17; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Stress, Psychological
Keywords: Psychology, Educational [F02.784.629]
MeSH Terms: conditions — Stress, Psychological | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: stress, psychological — students respond to questionnaires

SUMMARY:
Education is a process of human development for quality of life. Nurse anesthetist students in 1-year training program have to face occasional stress perioperatively such as long and unpredictable working hours, exposure to chemical and radiation hazards, or the occurrence of unexpected death, particularly when a given patient was previously healthy. This can sometimes prove frustrating and may lead to unsafe practices. Students with mild to moderate stress, act as achievement motive, driving them to succeed their goals in learning. However, anyone with severe stress often fails in his or her study. If learners face tension during their education and they are not able to solve it instantaneously; the stress becomes a vicious matter.

DETAILED DESCRIPTION:
Education is a process of human development for quality of life. It helps people to create ideas, judgement, problem solving or working ability with competency at their full strength. Currently, people are more demanding, lawyers more litigious, and insurance companies less willing to pay. In addition, hospital directors are trying to improve their management efficiency. As a result, doctors and nurses have to work harder. Sadly, the prevalence of burnout is higher among employees who deal with patients.

Anesthesia personnel have been at the forefront of the patient safety movement. They must be reliable and skilled at communicating with surgeons, operating room (OR) nurses, and ancillary workers. As a result, anesthetists have to maintain their physical, mental health, and special sensory capabilities.

Nurse anesthetist students in 1-year training program have to deal with stressful situation days and nights. The curriculum covering theoretical and practical learning in operating theater yields cumbersome atmosphere since medical errors have become a crucial society and professional issue. Inevitably, they face occasional stress perioperatively such as long and unpredictable working hours, exposure to chemical and radiation hazards, or the occurrence of unexpected death, particularly when a given patient was previously healthy. This can sometimes prove frustrating and may lead to unsafe practices.

Stress is a phenomenon that can happen to people in general. Students with mild to moderate stress, act as achievement motive, driving them to succeed their goals in learning. However, anyone with severe stress often fails in his or her study. If learners face tension during their education and they are not able to solve it instantaneously; the stress becomes a vicious matter that yields poor learning outcomes or even expel them from school. Consequently, stress may lead to some psychological problems. Stress in graduate students concerns to many influencing factors either to demean the situation or to diminish it. The stress-related factors are 1) studying: learning difficulties, daily rounds organization, exam preparation, and unfamiliar working circumstances 2) relationships: family members, instructors, consultants, friends, and colleagues 3) playing role: adult learning, conflict of interests in finance, physical or mental status. The previous studies revealed that these factors had evil effects on students tremendously.

As a result, investigators would like to study the stress-related factors in nurse anesthetist students during their learning program.

ELIGIBILITY:
Inclusion Criteria:

* voluntary, nurse anesthetist students without any honorarium

Exclusion Criteria:

* nurse anesthetist students can withdraw from the project at any time

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: nurse anesthetist students
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with stress as assessed by the specific tests | 1 year
  stress score

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Shayakul, M.D., Study Chair — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No